CLINICAL TRIAL: NCT06183918
Title: Appropriate Dose Of Tranexamic Acid In The Topical Treatment Of Anterior Epistaxis, 500mg Vs 1000mg; A Double-Blinded Randomized Controlled Trial
Brief Title: Tranexamic Acid Dosage for Topical Treatment of Anterior Epistaxis
Acronym: Tranexamicacid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cuneyt Arikan, Principal Investigator, Izmir Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IzmirATRH
Record Dates: First submitted 2023-07-27; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Anterior Epistaxis; Tranexamic Acid
Keywords: Anterior epistaxis; Tranexamic acid; Topical treatment; Emergency medicine
MeSH Terms: interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This randomized, double-blinded, phase-4 study. 3 different materials used to soak the gauze in nasal packing with gauze application, which is a treatment method for anterior epistaxis, were compared in terms of their superiority. First, those who met the study criteria and accepted to participate in the study and whose written consent was obtained were assigned to one of the treatment groups according to the next randomization number. Treatment groups were determined as;
  1. Group: Gauze soaked with 1000 mg TXA-topical
  2. Group: Gauze soaked with 500 mg TXA + 5 cc saline -topical
  3. Group: Gauze soaked with 10 cc of saline-topical.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The research products, saline and tranexamic acid ampoules containing 250 mg/2.5 ml of injectable solution, both in colorless, odorless, clean, and clear liquid form. The medications and medical supplies (gauze soaked with saline and TXA) to be used in the treatment according to the randomization number were prepared by a physician and a nurse working in the emergency room that were informed about the research priorly. Blindness was ensured by filling all groups to a 10 cc volume with saline. The prepared anterior nasal packing and medication administration were performed blindly by another emergency physician. Pressure was applied to both sides of the nose wings during the application for 10 minutes. Another researcher, who was not responsible for the preparation and administration of the medication, recorded the data in the Case Report Form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Group (Active Comparator): Gauze soaked with 1000 mg TXA-topical
  Interventions: Drug: Tranexamic acid
- 2. Group (Active Comparator): Gauze soaked with 500 mg TXA + 5 cc saline -topical
  Interventions: Drug: Tranexamic acid
- 3. Group (Active Comparator): Gauze soaked with 10 cc of saline-topical.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Tranexamic acid — 1. Group: Gauze soaked with 1000 mg TXA-topical
  2. Group: Gauze soaked with 500 mg TXA + 5 cc saline -topical The prepared anterior nasal packing and medication administration were performed. Pressure was applied to both sides of the nose wings during the application for 10 minutes. It was checked whether the bleeding continued at the 5th and 10th minutes after anterior nasal packing and medication administration.
  Arms: 1. Group; 2. Group
Other: Saline — 3. Group: Gauze soaked with 10 cc of saline-topical. The prepared anterior nasal packing and medication administration were performed. Pressure was applied to both sides of the nose wings during the application for 10 minutes. It was checked whether the bleeding continued at the 5th and 10th minutes after anterior nasal packing and medication administration.
  Arms: 3. Group

SUMMARY:
Patients with epistaxis usually apply to the emergency department for initial treatment. According to recent research, tranexamic acid is effective in the treatment of epistaxis. The research compare the therapeutic superiority of saline with 500 and 1000 mg doses of topical tranexamic acid in the treatment of anterior epistaxis. The design of the phase 4 clinical trial was randomized controlled double-blind. A total of 152 cases in 3 groups were included in the study. Group 1 was treated with 1000 mg of tranexamic acid, group 2 with 500 mg of tranexamic acid, and group 3 with saline. The primary outcome of the study was bleeding control at the 5th and 10th minutes. Secondary outcomes were determined as the need for salvage therapy, recurrent bleeding within 24 hours, the presence of side effects, and the need for otorhinolaryngology consultation.

DETAILED DESCRIPTION:
This randomized, double-blinded, phase-4 study was conducted in a single center between July and December 2022.

Among the patients aged 18 years and older who applied to the emergency department with epistaxis that accepted to participate in the study and could give written consent, patients with posterior epistaxis, with a history of nose or pharynx surgery in the last 3 months, with facial and head trauma, with unstable vital signs, patients who applied for the second time with a recurrent bleeding, patients with a history of allergy to TXA, patients with subarachnoid hemorrhage, patients with coagulation disorders such as hemophilia, hereditary telangiectasia, von Willebrand disease, etc., patients with thromboembolic disease, history of convulsions or intracerebral processes, and those who were pregnant or lactating, and who wished to withdraw from the study at any stage of the study were excluded from the study. 152 patients who did not meet the exclusion criteria were included in the study.

In this study, 3 different materials used to soak the gauze in nasal packing with gauze application, which is a treatment method for anterior epistaxis, were compared in terms of their superiority. Physicians and nurses participating in the study were given a total of 2 hours of theoretical and practical training on the design of the study and nasal packing application before the study. First, those who met the study criteria and accepted to participate in the study and whose written consent was obtained were assigned to one of the treatment groups according to the next randomization number. Treatment groups were determined as;

1. Group: Gauze soaked with 1000 mg TXA-topical
2. Group: Gauze soaked with 500 mg TXA + 5 cc saline -topical
3. Group: Gauze soaked with 10 cc of saline-topical. The research products, saline and tranexamic acid ampoules containing 250 mg/2.5 ml of injectable solution, both in colorless, odorless, clean, and clear liquid form. The medications and medical supplies (gauze soaked with saline and TXA) to be used in the treatment according to the randomization number were prepared by a physician and a nurse working in the emergency room that were informed about the research priorly. Blindness was ensured by filling all groups to a 10 cc volume with saline. The prepared ANP and medication administration were performed blindly by another emergency physician. Pressure was applied to both sides of the nose wings during the application for 10 minutes. Another researcher, who was not responsible for the preparation and administration of the medication, recorded the data in the Case Report Form (CRF). It was checked whether the bleeding continued at the 5th and 10th minutes after ANP and medication administration. In cases of bleeding lasting longer than ten minutes, one of the standard treatments used in epistaxis treatment (Sponge-shaped nasal tampon or inflatable balloon-shaped nasal tampon) was applied as salvage therapy, and otorhinolaryngology consultation was requested when necessary. In addition, patients were followed up for at least 1 hour in terms of possible side effects. Demographic data (age, gender), vital signs, use of anticoagulant and/or antiplatelet drugs, hemoglobin (Hgb), platelet (Plt), and International Normalized Ratio (INR) values of the cases, data of the applied procedure (5th and 10th minute bleeding control, necessity of salvage therapy), treatment-related side effects (administration site reaction, rash, rash, itching, erythema, urticaria, hives, chest pain, dyspnea, nausea, vomiting, blackout, headache, dizziness), the need for otorhinolaryngology consultation, and whether recurrency developed within 24 hours was recorded in the CRF. Participants were advised to inform the principal investigator by telephone if recurrent bleeding occurs within 24 hours and to apply to the emergency department again in case of recurrent and/or prolonged bleeding.

The primary outcome of the study was bleeding control at the 5th and 10th minutes. Secondary outcomes were determined as the need for salvage therapy, recurrent bleeding within 24 hours, the presence of side effects, and the need for otorhinolaryngology consultation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Those who applied to the emergency department with the complaint of nosebleeds
* Those who agreed to participate in the study by giving written consent

Exclusion Criteria:

* posterior epistaxis
* history of nose or pharynx surgery in the last 3 months,
* facial and head trauma,
* unstable vital signs,
* who applied for the second time with a recurrent bleeding
* history of allergy to TXA,
* subarachnoid hemorrhage,
* coagulation disorders such as hemophilia, hereditary telangiectasia, von Willebrand disease, etc.
* thromboembolic disease
* history of convulsions
* intracerebral processes
* pregnant or lactating
* who wished to withdraw from the study at any stage of the study

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Number of cases whose nosebleeds were completely stopped | 5th and 10th minutes
  Number of cases in which nosebleeds were completely stopped at the 5th and 10th minutes

SECONDARY OUTCOMES:
Need for salvage therapy | After 10 minutes
  Cases whose bleeding cannot be controlled and need additional treatment
The presence of side effects | 1 hour
  Treatment-related side effects (administration site reaction, rash, rash, itching, erythema, urticaria, hives, chest pain, dyspnea, nausea, vomiting, blackout, headache, dizziness)
Need for otorhinolaryngology consultation | After 1 hour
  Number of cases whose bleeding cannot be controlled despite salvage treatment or for which otorhinolaryngology consultation is requested for another reason
Recurrent bleeding within 24 hours | 24 hours
  Number of cases with recurrent bleeding within 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk 'Training and Research Hospital, Izmir, Basın Sitesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data of the research will be shared upon the request of the competent health authorities.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years